CLINICAL TRIAL: NCT00394537
Title: Labetalol to Prevent Hypertension and Tachycardia During Fiberoptic Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3997
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-05

CONDITIONS: Bronchoscopy
MeSH Terms: interventions — Labetalol

INTERVENTIONS:
Drug: Labetalol 10mg iv

SUMMARY:
Passing a bronchoscope through the airways frequently causes a stress response even though patients are sedated. This stress response is usually an increase in pulse and blood pressure, which may have undesirable effects on the heart and circulation.

We plan to give patients labetalol (a beta blocker which reduces pulse and blood pressure) in addition to normal sedation, to patients undergoing bronchoscopy in our department.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old undergo fiberoptic bronchoscopy in our unit

Exclusion Criteria:

* inability or refusal to give informed consent
* bronchoscopy through an artificial airway
* intolerance or allergy to the study drug
* bradycardia (HR<60/min) or hypotension (systolic BP <100) at screening
* pregnancy,
* concomitant treatment with diltiazem or verapamil
* intention to use propofol as the sedative agent for bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate
Systolic Blood Pressure
Diastolic Blood Pressure
Rate pressure product (HR*SBP/100)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kramer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Fox BD, Krylov Y, Leon P, Ben-Zvi I, Peled N, Shitrit D, Kramer MR. Benzodiazepine and opioid sedation attenuate the sympathetic response to fiberoptic bronchoscopy. Prophylactic labetalol gave no additional benefit. Results of a randomized double-blind placebo-controlled study. Respir Med. 2008 Jul;102(7):978-83. doi: 10.1016/j.rmed.2008.02.011. Epub 2008 Apr 3. PMID 18394874